CLINICAL TRIAL: NCT05016024
Title: A Randomized, Cross-over, Placebo-Controlled, Double-Blind Clinical Trial on the Efficacy and Safety of Oral Administration of a Molecular Complex of Resins, Polysaccharides and Polyphenols in the Treatment of Irritable Bowel Syndrome
Brief Title: Administration of a Molecular Complex of Resins, Polysaccharides and Polyphenols in Irritable Bowel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: IQVIA RDS Inc. (Industry); IQVIA Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABO-COL-01/21
Record Dates: First submitted 2021-05-25; First posted 2021-08-23 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Colilen IBS; Abdominal Pain; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: Run in period: 2 weeks First Period: two months of treatment with Colilen IBS or Placebo, based on the randomization at Baseline visit Wash out period:3 weeks Second Period: two months of treatment with Colilen IBS or Placebo, based on the randomization at Baseline visit
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colilen IBS + Placebo (Other): First Period: Colilen IBS Second Period: Placebo
  Interventions: Device: Colilen IBS; Other: Placebo
- Placebo + Colilen IBS (Other): First Period: Placebo Second Period: Colilen IBS
  Interventions: Device: Colilen IBS; Other: Placebo

INTERVENTIONS:
Device: Colilen IBS — Patients will take Colilen IBS in First or Second Period
Other: Placebo — Patients will take PlaceboS in First or Second Period

SUMMARY:
This study is aimed to investigate the efficacy and safety of Colilen IBS, a Medical Device made of natural substances, even when taken in addition to other therapies, for the treatment of Irritable Bowel Syndrome.

DETAILED DESCRIPTION:
This is a Post Market, randomized, double blind, cross-over clinical evaluation that will be conducted in 66 patients with diagnosis of Irritable Bowel Syndrome according to Rome IV criteria. As this is a cross-over clinical investigation, each eligible patient will take both the products under investigation, Colilen IBS and its Placebo.

After a 2-week run-in period, at Baseline visit each patient included in the study will be randomly assigned to one of the two treatment sequences (i.e., Sequence AB and Sequence BA), for a 16-week total sequential treatment period (8 weeks for each of the 2 treatment periods) first with verum Colilen IBS and then with its Placebo, or vice versa. A wash out period (3 weeks) is forecast between the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients aged 18 to 75 years (inclusive);
* 2. Diagnosis of IBS according to ROME IV criteria (Appendix 3);
* 3. Abdominal pain score ≥ 4 on a 11-point NRS, on at least 2 days of the 14 days prior to the baseline visit and on at least 2 days of the last 14 days of the washout period, and pain score not > 8 in more than 7 days of each of the two above-mentioned periods;
* 4. Signed Informed Consent;
* 5. Patients' ability to comply with the study procedures;
* 6. Stable diet in the two months prior to the screening visit;
* 7. *Negative colonoscopy, defined as the absence of clinically relevant changes or of changes nonetheless relevant in relation to study participation risk, performed during the run-in period, unless:

  * a colonoscopy was performed within the previous 5 years and was negative as intended above, or, if more than one was performed within the previous 5 years, the last being negative as intended above;
  * the symptoms, if any, for which the last colonoscopy was performed, have remained unchanged;
* 8. Postmenopausal female patients, i.e., females who have not had a menstrual period for at least 12 months or women who have undergone surgical sterilisation (tubal ligation or ovary removal). If not, women of childbearing potential must follow reliable contraceptive treatment.

  * Inclusion criteria applicable only for patients > 50 years of age

Exclusion Criteria:

* 1. Patients taking treatments that may significantly affect the efficacy outcomes measures, such as: probiotics and prebiotics (unless contained in milk-derived foods such as yogurt and cheese); drugs with adsorbent/sequestrant properties such as diosmectite; 5-HT3 receptor antagonist drugs, e.g. ondasetron; drugs that modify gastro-intestinal motility, e.g. "final" anti-cholinergic agents such as loperamide, or cholinergic agents; laxatives and faecal softeners) unless they have been taken at a stable dose for at least four weeks prior to the screening visit.
* 2. Patients taking tricyclic antidepressants within six months prior to the screening visit;
* 3. Patients taking opioid-containing analgesics within one month prior to the screening visit;
* 4. Patients taking antibiotics within one month prior to the screening visit;
* 5. Patients with relevant organic, systemic or metabolic disease, or laboratory changes, that are deemed significant based on specific ranges of normality;
* 6. Patients with organic bowel diseases;
* 7. Patients with unstable psychiatric conditions;
* 8. Patients who have undergone major abdominal surgery, except appendectomy;
* 9. Known hypersensitivity to one or more of the components of the products.
* 10.Women with known or planned pregnancy or breastfeeding;
* 11.Patients with malignancies of any type, or with a history of prior malignancies, except for patients with a history of extra-intestinal malignancies that have been surgically removed and have not relapsed within the five years prior to participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline after treatment in: Symptom intensity sum score (flatulence/meteorism, feeling of turgidity or fullness, feeling of incomplete evacuation, changes in bowel habit) | End of treatment (up to 5 months)
  The endpoint will be assessed through a 4-point Likert scale (minimum sum score: 0; maximun sum score:12).
Change from baseline after treatment in: Abdominal pain intensity sum score on an 11-point numeric rating scale, NRS (from 0 to 10). | End of treatment (up to 5 months)
  The endpoint will be assessed through an 11-point numeric rating scale (NRS, from 0 to 10)

SECONDARY OUTCOMES:
Change from baseline in IBS-SSS (symptom severity score). | End of treatment (up to 5 months)
  Irritable Bowel Syndrome-Severity Scored System (IBS-SSS) questionnaire. The maximum achievable score is 500. Mild, moderate and severe cases were indicated by scores of 75 to 175, 175 to 300 and > 300 respectively.
Change of adequate overall symptom relief after treatment, defined by a score of at least 3 on a 7-point Likert scale of weekly relief, in at least 50% of treatment weeks: | End of treatment (up to 5 months)
  7-point Likert Scale" Possible answers: 1, very relieved; 2, relieved; 3, somewhat relieved; 4, unchanged; 5, slightly worsened; 6, worsened; 7, much worsened (7-point Likert Scale).
Time to adequate overall relief of IBS symptoms. | End of treatment (up to 5 months)
  Score of a 7-point Likert scale 7-point Likert Scale" Possible answers: 1, very relieved; 2, relieved; 3, somewhat relieved; 4, unchanged; 5, slightly worsened; 6, worsened; 7, much worsened
Change from baseline after treatment in: o Severity score of each of the individual symptoms included in the IBS-SSS (sub-scores), assessed by a NRS from 0 to 100; | End of treatment (up to 5 months)
  IBS-SSS (Syndrome Severity Scoring) questionnaire sub score
Change from baseline after treatment in: Quality of life as assessed by IBS-QoL (Quality of Life). | End of treatment (up to 5 months)
  IBS-QoL Questionnaire
Change from baseline after treatment in the different clinical subgroups according to the presence of prevalent bowel changes, including: Bowel movement frequency; | End of treatment (up to 5 months)
  Daily diary
Change from baseline after treatment in the different clinical subgroups according to the presence of prevalent bowel changes, including: Stool consistency according to Bristol stool form scale (BSFS); | End of treatment (up to 5 months)
  BSFS (Bristol Stool Form Scale)
Change from baseline after treatment in the different clinical subgroups according to the presence of prevalent bowel changes, including: IBS-SSS NRS sub-score of bowel movement satisfaction. | End of treatment (up to 5 months)
  IBS-SSS (Syndrome Severity Scoring) questionnaire
Change from baseline halfway through treatment in: IBS-SSS (Syndrome Severity Scoring) symptom severity score; | 1 month
  IBS-SSS (Syndrome Severity Scoring) questionnaire
Change from baseline halfway through treatment in: Severity score of each of the individual symptoms included in the IBS-SSS (sub-scores), assessed by a NRS from 0 to 100; | 1 month
  IBS-SSS (Syndrome Severity Scoring) questionnaire
Change from baseline halfway through treatment in: Bowel movement frequency in the clinical subgroup with a predominating bowel movement change; | 1 month
  Daily diary
Change from baseline halfway through treatment in: Stool consistency according to the Bristol scale in the clinical subtype with a predominating bowel movement change. | 1 month
  BSFS (Bristol Stool Form Scale)
Change from baseline halfway through treatment in: IBS-SSS NRS sub-score of bowel movement satisfaction in the clinical subtype with no predominating bowel changes, i.e., IBS-M (mixed) and IBS-U (unclassified). | 1 month
  IBS-SSS (Syndrome Severity Scoring) questionnaire
Change from baseline after treatment in the type and number of concomitant therapies taken for IBS symptoms. | End of treatment (up to 5 months)
  number of concomitant therapies
Incidence of AEs during study treatment | End of treatment (up to 5 months)
  Incidence and type of adverse events (AEs) and serious adverse events (SAEs) reported during study treatment.
  Safety will be assessed on the basis of all AEs experienced during study treatment. Furthermore, change from baseline in safety laboratory parameters and clinical examination findings (including measurement of anthropometric parameters and vital signs such as systolic/diastolic blood pressure, pulse, weight) will be assessed.

CONTACTS AND LOCATIONS:
Locations (7):
- Klinische Forschung Karlsruhe GmbH, Karlsruhe, Germany
- Italy (6):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Ospedale SS. Annunziata, Chieti
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Policlinico Universitario A. Gemelli, Rome